CLINICAL TRIAL: NCT00131326
Title: A Study of the Safety and Efficacy of Synvisc and Depo-Medrol in Patients With Osteoarthritis of the Hip
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYNV-004-02
Record Dates: First submitted 2005-08-17; First posted 2005-08-18 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Osteoarthritis, Hip; Musculoskeletal Diseases
Keywords: osteoarthritis of the hip; Musculoskeletal Diseases
MeSH Terms: conditions — Osteoarthritis, Hip; Musculoskeletal Diseases

INTERVENTIONS:
Device: Synvisc (hylan G-F 20)

SUMMARY:
This is a clinical study to investigate the safety and efficacy of Synvisc and Depo-Medrol in treating patients with osteoarthritis (OA) of the hip.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic osteoarthritis pain of hip

Exclusion Criteria:

* Patients with current or prior conditions or treatment that would impede measurement of efficacy and safety

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-11; Study Completion 2006-04

PRIMARY OUTCOMES:
Pain relief

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (32):
- United States (32):
  - Alabama Clinical Therapeutics, Birmingham, Alabama
  - John Higginbotham, MD Sports Medicine, Huntsville, Alabama
  - Affiliated Orthopedic Specialists, Scottsdale, Arizona
  - Arkansas Orthopaedic Specialists, Little Rock, Arkansas
  - Cedars-Sinai Orthopedic Center, Los Angeles, California
  - Jackson Arthritis Center, Oakland, California
  - Orthopedic Medical Group, San Diego, California
  - Orthopedic Specialists of Tamp Bay, P.A., Clearwater, Florida
  - Orthopedic Institute at Mercy Hospital, Miami, Florida
  - Hughston Sports Medicine Foundation, Columbus, Georgia
  - Idaho Arthritis & Osteoporosis Center, Meridian, Idaho
  - Northwestern Orthopaedic Institute, Chicago, Illinois
  - Illinois Bone and Joint Institute, Ltd., Morton Grove, Illinois
  - David S. Tearse, MD (Private Practice), Cedar Rapids, Iowa
  - Kansas City Orthopedic Institute, Leawood, Kansas
  - Bluegrass Orthopaedics, Lexington, Kentucky
  - Orthopedic Specialists of Louisiana, Shreveport, Louisiana
  - Maryland General Hospital, Baltimore, Maryland
  - Family Orthopedic Associates, Flint, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - UMDNJ-RWJ University Orthopedic Group, New Brunswick, New Jersey
  - Hospital for Special Surgery, New York, New York
  - Health Research Institute, Oklahoma City, Oklahoma
  - Orthopedic Center for Joint Replacement & Sports Medicine, Grants Pass, Oregon
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Lancaster Orthopedic Group, Lancaster, Pennsylvania
  - Allegheny Orthopedic Associates, Pittsburgh, Pennsylvania
  - Conway Medical Center, Conway, South Carolina
  - Chattanooga Center for Sports, Chattanooga, Tennessee
  - Gurdev Gill, MD (Private Practice), Lubbock, Texas
  - Carilion Bone and Joint Center, Vinton Orthopedic Surgery, Vinton, Virginia
  - Arthritis Northwest, Seattle, Washington

REFERENCES:
- [Background] Spitzer AI, Bockow BI, Brander VA, Yates JW, MacCarter DK, Gudger GK, Haller S, Lake SL, Magilavy DB. Hylan G-F 20 improves hip osteoarthritis: a prospective, randomized study. Phys Sportsmed. 2010 Jun;38(2):35-47. doi: 10.3810/psm.2010.06.1781. PMID 20631462